CLINICAL TRIAL: NCT07205536
Title: A Clinical Study on the Safety and Efficacy of Mecapegfilgrastim in Preventing Myelosuppression Induced by Concurrent Chemoradiotherapy for Thoracic Malignancies
Brief Title: Clinical Study of Thiopegfilgrastim for Preventing Bone Marrow Suppression in Thoracic Tumor Chemoradiotherapy
Acronym: ANC-IIT-004
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-K299-01
Record Dates: First submitted 2025-09-18; First posted 2025-10-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-08

CONDITIONS: Myelosuppression; Thoracic Neoplasms; Chemoradiotherapy
Keywords: Neutropenia; Febrile neutropenia
MeSH Terms: conditions — Thoracic Neoplasms; Neutropenia; Febrile Neutropenia | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral or short-acting granulocyte-stimulating agents (Active Comparator): When the neutrophil count falls below 1.5 × 10⁹/L, the investigator will discuss with the patient whether to initiate standard granulocyte-boosting therapy such as leucogen tablets.
  Interventions: Drug: Oral or short-acting granulocyte-stimulating agents
- Mecapegfilgrastim injection (Experimental): Administer a single subcutaneous injection of mecapegfilgrastim 24 hours after the end of each chemotherapy cycle. The recommended dose is a fixed 6 mg, or individualised dosing at 100 μg/kg based on patient body weight.
  Interventions: Drug: Mecapegfilgrastim injection

INTERVENTIONS:
Drug: Mecapegfilgrastim injection — After enrollment, a single subcutaneous dose of mecapegfilgrastim should be administered 24 hours following completion of each chemotherapy cycle. The recommended dose is a fixed 6 mg, or an individualized 100 μg/kg based on the patient's body weight. If neutrophil counts remain below 0.5 × 10⁹/L for more than 24 hours after mecapegfilgrastim administration, short-acting G-CSF may be used as rescue therapy at the investigator's discretion until neutrophil levels return to normal.
  Arms: Mecapegfilgrastim injection
Drug: Oral or short-acting granulocyte-stimulating agents — In the first cycle after enrollment, patients will be followed for changes in neutrophil counts. Should the neutrophil level fall below 1.5 × 10⁹/L, the investigator may, based on clinical judgment, decide whether to intervene with leucogen tablets or other granulocyte-boosting agents. If the count remains below 1.0 × 10⁹/L, short-acting G-CSF may be administered as a rescue therapy.
  Arms: Oral or short-acting granulocyte-stimulating agents

SUMMARY:
This is a prospective observational study designed to observe and evaluate the safety and efficacy of mecapegfilgrastim in the treatment of moderate-to-severe myelosuppression associated with concurrent chemoradiotherapy. The project will provide more robust evidence-based medical support for the use of long-acting granulocyte-stimulating agents in patients undergoing concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
Group 1: Monitor the changes in neutrophil levels during the first follow-up cycle after enrollment in this study. When the neutrophil level falls below 1.5×10⁹/L, the investigator will communicate with the patient to determine whether to use conventional leukocyte-increasing drugs such as Licorice tablets. If so, the patient will be assigned to Group 1.

Group 2: After enrollment in this study, the investigator will communicate with the patient to determine whether to use Sulfated PEG-Interferon injection to prevent and treat neutropenia. If so, 24 hours after the end of the chemotherapy cycle, the patient will receive a subcutaneous injection of Sulfated PEG-Interferon once. The recommended dose is a fixed dose of 6 mg per injection; or, based on the patient's weight, an individualized treatment dose of 100 μg/kg. The patient will then be assigned to Group 2.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years at the time of giving informed consent， both sexes eligible
* Histologically or cytologically confirmed thoracic tumor (esophageal or lung cancer)
* Investigator judges the patient suitable for treatment with mecapegfilgrastim injection or leucogen tablets
* Expected survival > 3 months
* Signed informed consent; willing and able to comply with protocol-mandated visits
* The patient is indicated for concurrent chemoradiotherapy and is currently/receiving or will receive a high-risk chemotherapy regimen for febrile neutropenia (FN risk ≥20%), or is currently/receiving or will receive an intermediate-risk chemotherapy regimen for FN (FN risk 10%~20%) with additional FN risk factors.

Exclusion Criteria:

* Pregnant or lactating women
* Known hypersensitivity to mecapegfilgrastim, pegylated or non-pegylated rhG-CSF, or any E. coli-derived product
* Any severe comorbidity that, in the investigator's opinion, compromises patient safety or ability to complete the study
* Any other condition that, in the investigator's judgment, could interfere with study conduct or interpretation of results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of hematologic toxicity | Day 7,Day 14
  Hematologic toxicity, assessed by CBC performed 1 day before chemotherapy and on days 7 and 14 post-chemotherapy; CBC may be done at an external facility.

SECONDARY OUTCOMES:
The incidence of non-hematologic toxicity | Day 1, Day 7, and Day 14 of the first and second anti-tumor treatment cycles, and Day 30 after the completion of radiotherapy.
  Secondary Outcome Measures: Non-hematologic toxicity On Day 1 of cycles 1 and 2: vital signs, complete blood count, urinalysis, stool routine, serum chemistry, coagulation panel, and 12-lead ECG.
  On Days 7 and 14 of cycles 1 and 2: repeat complete blood count only. All patient-reported adverse events are captured through 30 days after completion of radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided